CLINICAL TRIAL: NCT03887806
Title: Efficacy Cost Analysis: Retrospective Study on the REMOTEV Study's Ancillary Data
Brief Title: Cost Effectiveness Analysis of an Ancillary Study of the REMOTEV Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7158
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Venous Thromboembolic Disease
Keywords: Venous; Thromboembolic; Direct Oral Anticoagulants; AOD; Cost analysis; REMOTEV; AVK; Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The implications of the medico-economic impact are essential in the choice of first-line therapists. The economic impact is an important criterion to recommend the privileged use of Direct Oral Anticoagulants (AOD) in first intention.

ELIGIBILITY:
Inclusion criteria

* Major patient whose age is ≥18 years
* Patient with a diagnosis of MTEV: pulmonary embolism or deep vein thrombosis diagnosed by the diagnostic reference methods according to the recommendations
* Major patient included in the REMOTEV registry
* Patient having accepted that his data recorded in the REMOTEV register be re-used for research and publication purposes

Criteria of non-inclusion

* Refusal to participate in the REMOTEV register
* Patient who refused to have his data reused for research and publication purposes
* Pregnant woman
* Subjects under safeguard of justice Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a diagnosis of MTEV: pulmonary embolism or deep vein thrombosis diagnosed by the diagnostic reference methods according to the recommendations
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-03-20 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness analysis between 2 therapeutic strategies, Direct Oral Anticoagulants (Rivaroxaban) versus standard anticoagulant (AVK) | The period from November 1st, 2013 to July 01, 2015 will be examined
  Cost-effectiveness analysis between 2 therapeutic strategies: The costs related to each strategy are calculated taking into account the direct and indirect costs.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique STEPHAN, MD, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service Des Maladies Vasculaires - Hta - Nhc, Strasbourg, France